CLINICAL TRIAL: NCT00925366
Title: Comparative Performances of CT-arthrography, MRI and MR-arthrography in the Preoperative Assessment of the Rotator Cuff Tendon Tears, Surgical Observations Being Used as a Standard.
Brief Title: Which is the Most Reliable Radiologic Examination for the Diagnosis of Rotator Cuff Tendon Tear?
Acronym: COIFFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department of Clinical Research of Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P020909
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-06

CONDITIONS: Shoulder; Rotator Cuff Disease
Keywords: Shoulder; MRI; MR arthrography; CT arthrography; Rotator cuff tear; Arthroscopy
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shoulder rotator cuff tear (Other): Shoulder rotator cuff tear
  Interventions: Other: Imaging Procedure

INTERVENTIONS:
Other: Imaging Procedure — CT Arthroscopy of the Shoulder - MR Arthroscopy of the Shoulder - MR of the shoulder

SUMMARY:
At this point in time the approach to the diagnosis of rotator cuff tendon tears is not consensual. The French surgeons, considering they have a good experience of this method, preferably use a shoulder CT-arthrography. Whereas in the United States surgeons rather rely on MRI or MR-arthrography of the shoulder. However, nobody can say which of these three examinations is most precise and gives the best information. We proposed to carry out the three examinations at the same time in a large number of patients who needed to be operated for a rotator cuff tendon tear and then to compare the results of each of these examinations with the operative observations.

DETAILED DESCRIPTION:
Rotator cuff tendon tear is the principal pathology of the shoulder. These degenerative tendon lesions are due to normal ageing. True complete asymptomatic tears are even quite frequently noted in old subjects. However, they can be very invalidating. The majority of these degenerative lesions are treated medically. In a limited number of cases, a surgical treatment aimed at reducing a mechanical conflict and/or repair the tendons is necessary.

The indication for a surgical treatment is based on the clinical evaluation and the radiological assessment. The radiological assessment is essential to confirm the tears but also to evaluate their extent. The type of surgery depends on this anatomic and radiologic assessment. It is thus possible, in the event of small complete tear, to make a simple tendon suture or a transosseous reinsertion. On the other hand, in the event of a large tear with tendon retraction, muscular flap reconstruction is needed.

The preoperative radiological assessment is based on different radiological examinations, exploring the tendons. In the United States, MRI is mainly used in this case. In France, it is CT-arthrography which is regarded as the standard of care because the high contrast resolution of the images obtained and their reliability appear to be higher than those of MRI. The articular puncture necessary to perform this examination is not regarded in our country as an obstacle. The MR-arthrography, which consists in injecting into the joint of very low concentration of gadolinium, makes it possible to obtain an arthrographic effect in MRI. This examination gives images with an excellent contrast. It is already very widespread in the USA. In France, we have an increasingly large experience of it, but still limited.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is > to 18 years
* Patient presenting a clinical suspicion of rotator cuff tear
* Obtaining the enlightened consent of the patient

Exclusion Criteria:

* Patient having refused to sign his consent
* Patient whose age is < to 18 years.
* Patient with capsulitis
* Patient presenting history of allergy.
* Patient presenting an anticoagulant or salicylated treatment which can not be interrupted.
* Pregnant woman.
* Patient with a contra-indication to MRI.
* Patient with a psychiatric pathology preventing a clinical evaluation.
* Patient with contra-indication (cutaneous or different) to the intra-articular injection.
* Patient with a history of non degenerative pathology in the same shoulder (inflammatory disease, serious infection, tumor…) or with past intervention on the same shoulder.
* Surgery contra-indication (cardiac failure, respiratory…)
* Patient without health coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-09; Primary Completion 2007-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To determine which of the 3 radiological examinations, MRI, MR-arthrography and CT-arthrography, is the best in term of sensitivity, specificity and predictive value, in the preoperative assessment of rotator cuff tears. | 6 months

SECONDARY OUTCOMES:
To improve our knowledge of the radiological aspect of degenerative lesions of rotator cuff tendon thanks to clinical, radiological and surgical confrontations | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis Laredo, Pr, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital LARIBOISIERE Service de Radiologie Ostéo-Articulaire, Paris, France